CLINICAL TRIAL: NCT05092035
Title: Recognition of Early Pulmonary Structural Changes by Using Real-time High Fidelity Expiratory CO2 Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ID 7684
Record Dates: First submitted 2021-08-04; First posted 2021-10-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: COPD; ILD
Keywords: structural pulmonary changes; High fidelity analysis of expiratory CO2 flow
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: 3 Groups, two control Groups (smokers and non-smokers), one COPD group, one ILD group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- COPD patients (Other): COPD patients
  Interventions: Diagnostic Test: single high-fidelity expiratory CO2 analysis
- ILD patients (Other): ILD patients
  Interventions: Diagnostic Test: single high-fidelity expiratory CO2 analysis
- non-smoker controls (Other): non-smoker controls
  Interventions: Diagnostic Test: single high-fidelity expiratory CO2 analysis
- smoker controls (Other): smoker controls
  Interventions: Diagnostic Test: single high-fidelity expiratory CO2 analysis

INTERVENTIONS:
Diagnostic Test: single high-fidelity expiratory CO2 analysis — in addition to regular pulmonary function testing a real-time high-fidelity assessment of expiratory CO2 will be performed

SUMMARY:
In this study the investigators aim to detect and characterize structural airway and lung vessel changes due to COPD or ILD as assessed by real-time high fidelity expiratory CO2 analysis. The long-term goal is to detect pulmonary structural changes in a stage, when variables of currently used standard methods (e.g. pulmonary function test) are not yet altered.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the fourth leading cause of death worldwide and is responsible for over 6% of all-cause mortality. Due to aging societies and exposure to risk factors, increasing prevalence is expected in the following years. Cigarette smoking is the most important risk factor for COPD, but also non-smokers may develop the disease. Although COPD is primarily seen as obstructive airway disease, it may also affect the lung parenchyma, the lung vessels, the systemic vessels, the heart and other organs. Therefore, COPD may be seen as a "pulmonary component of a systemic disease ". According to recent evidence patients with COPD and relevant lung vessel disease are at a higher risk to develop exacerbations and have worse prognosis. Usually, COPD patients suffer from a mild pulmonary hypertension, however some of them may present with a "pulmonal vascular phenotype" (PVP). Patients with PVP usually suffer from a relatively mild airway obstruction and are characterized by pathological changes in the small lung vessels, strongly elevated pulmonary vascular resistance, severely reduced diffusion capacity, normo- or hypocapnia, circulatory limitation of exercise capacity and a progressive right heart failure. Early recognition and therapy of COPD may stop further progression of the disease and the development of complications including changes in the small lung vessel.

Interstitial lung diseases (ILD) are characterized by structural changes in the lungs with fibrotic destruction and loss of alveolar tissue. Male gender and smoke exposure are frequent risk factors. At the time of diagnosis, patients are usually in an impaired physical condition suffering from severe symptoms and advanced functional limitation. In a subgroup of patients, a severe lung vessel disease is present further worsening prognosis. Although in the past few years major improvements in the therapy of some forms of ILD have been achieved, the available drugs are not curative. Their aim remains to slow down disease progression. Therefore, an early detection of ILDs may help to initiate targeted treatment on time and improve the prognosis of patients.

Structural pulmonary changes both due to COPD or ILD result in a loss of small airways and small lung vessels, which are not detectable with standard pulmonary function tests until 50% of the small airways disappeared. Although these changes may also take place due to physiological lung-aging, in smokers this effect is clearly accelerated. Diffusion capacity (DLCO) and the so-called Krogh factor (KCO) are sensible markers of early pulmonary structural changes. In addition, lung density as assessed by high-resolution CT-scan and analyzed by specific software represents a sensitive tool. Pulmonary vascular resistance (PVR) and pulmonary vascular compliance are sensitive parameters for the detection of pulmonary vascular changes.

Similar to DLCO, high fidelity analysis of expiratory CO2-flow measurement may allow a sensitive detection of structural pulmonary changes. The method has the advantage that no extrinsic gas is needed. The aim of this explorative pilot study is to investigate if high fidelity expiratory CO2-analysis is able to detect early pulmonary structural changes, even before it can be assessed by pulmonary function testing (e.g. FEV1 or vital capacity).

ELIGIBILITY:
Inclusion Criteria:

* all male and female patients older than 18 years who have COPD, ILD or are smokers and non smokers without pulmonary diseases.
* right heart catheterization performed due to to suspected pulmonary hypertension and further clinical investigation like echocardiography, lung function testing, 6-minute walk test, laboratory testing and blood gas analysis.
* written informed consent

Exclusion Criteria:

* contraindication for lung function testing
* acute life-threatening disease (including acute myocardiac infarction, pulmonary embolism, large aortic aneurysma, pneumothorax, opthalmic, brain, abdominal or thoracic surgery within the last 4 weeks, hemoptysis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
change in partial pressure of CO2 (in mmHg) during expiration | 1 day
  the change in real-time high-fidelity partial pressures of CO2 (in mmHg) during expiration will be compared among groups

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, Prof., Principal Investigator — Devision of Pulmonology, Medical University Hospital of Graz, Austria
Locations (1):
- Department of Internal Medicine, Pulmonology, Graz, Styria, Austria

REFERENCES:
- [Result] Singh D, Agusti A, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Criner GJ, Frith P, Halpin DMG, Han M, Lopez Varela MV, Martinez F, Montes de Oca M, Papi A, Pavord ID, Roche N, Sin DD, Stockley R, Vestbo J, Wedzicha JA, Vogelmeier C. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease: the GOLD science committee report 2019. Eur Respir J. 2019 May 18;53(5):1900164. doi: 10.1183/13993003.00164-2019. Print 2019 May. PMID 30846476
- [Result] Tanabe N, Vasilescu DM, McDonough JE, Kinose D, Suzuki M, Cooper JD, Pare PD, Hogg JC. Micro-Computed Tomography Comparison of Preterminal Bronchioles in Centrilobular and Panlobular Emphysema. Am J Respir Crit Care Med. 2017 Mar 1;195(5):630-638. doi: 10.1164/rccm.201602-0278OC. PMID 27611890
- [Result] McDonough JE, Yuan R, Suzuki M, Seyednejad N, Elliott WM, Sanchez PG, Wright AC, Gefter WB, Litzky L, Coxson HO, Pare PD, Sin DD, Pierce RA, Woods JC, McWilliams AM, Mayo JR, Lam SC, Cooper JD, Hogg JC. Small-airway obstruction and emphysema in chronic obstructive pulmonary disease. N Engl J Med. 2011 Oct 27;365(17):1567-75. doi: 10.1056/NEJMoa1106955. PMID 22029978
- [Result] Nathan SD, Barbera JA, Gaine SP, Harari S, Martinez FJ, Olschewski H, Olsson KM, Peacock AJ, Pepke-Zaba J, Provencher S, Weissmann N, Seeger W. Pulmonary hypertension in chronic lung disease and hypoxia. Eur Respir J. 2019 Jan 24;53(1):1801914. doi: 10.1183/13993003.01914-2018. Print 2019 Jan. PMID 30545980
- [Result] Kovacs G, Agusti A, Barbera JA, Celli B, Criner G, Humbert M, Sin DD, Voelkel N, Olschewski H. Pulmonary Vascular Involvement in Chronic Obstructive Pulmonary Disease. Is There a Pulmonary Vascular Phenotype? Am J Respir Crit Care Med. 2018 Oct 15;198(8):1000-1011. doi: 10.1164/rccm.201801-0095PP. No abstract available. PMID 29746142